CLINICAL TRIAL: NCT00641082
Title: A Double-Blind Randomized Clinical Trial Comparing the Safety and Antiviral Activity of 48-week Clevudine and Adefovir Dipivoxil in HBeAg(-) Chronic Hepatitis B With Compensated Liver Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLV-401
Record Dates: First submitted 2008-03-05; First posted 2008-03-21 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: HBeAg(-) Chronic Hepatitis B With Compensated Liver Function
MeSH Terms: interventions — clevudine; adefovir dipivoxil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Clevudine
  Interventions: Drug: Clevudine
- 2 (Active Comparator): Adefovir
  Interventions: Drug: Adefovir dipivoxil

INTERVENTIONS:
Drug: Clevudine — 30mg for 48 weeks
  Other Names: Levovir
  Arms: 1
Drug: Adefovir dipivoxil — 10mg for 48 weeks
  Other Names: Hepsera
  Arms: 2

SUMMARY:
A double-blind randomized, parallel, multicenter with 48 weeks of treatment period. The purpose of this study is to compare the safety and antiviral activity of 48-week Clevudine and Adefovir dipivoxil in HBeAg(-) Chronic Hepatitis B with compensated liver function.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 60
* Patient is documented to be HBsAg positive for > 6 months.
* Patient with compensated hepatic function.
* Nucleoside treatment-naÃ-ve subjects of either gender
* Patient is HBeAg negative. Patient is HBV DNA positive with DNA levels â‰¥ 1 x 10(5) copies/mL within 30 days of baseline.
* Patient has ALT levels which are in the range of 2 x ULN and < 10 X ULN
* Patient who has not a history of ascites, variceal hemorrhage or hepatic encephalopathy.

Exclusion Criteria

* Patient is currently receiving antiviral or corticosteroid therapy.
* Patients previously treated with lamivudine, adefovir, entecavir, telbivudine, clevudine, lobucavir, famciclovir or any other investigational nucleoside for HBV infection.
* Previous treatment with interferon must have ended at least 6 months prior to the screening visit.
* Treatment with nephrotoxic drugs, competitors of renal excretion, and/or hepatotoxic drugs within 2 months before study screening or during the study period
* Subjects who are currently participating in another investigational study or has been taking any investigational drug within the last 4 weeks prior to screening visit.
* Patient is coinfected with HCV, HDV or HIV.
* Patient with following clinical evidence

  * Decompensated liver cirrhosis (Child class B,C: CPT score 7) or hepatocellular carcinoma
  * Significant gastrointestinal, renal, bronchopulmonary, neurological, cardiovascular, oncologic or allergic disease
* Previous organ transplantation
* Patient has a clinically relevant history of abuse of alcohol or drugs.
* Patient is pregnant or breast-feeding.
* Patient is unwilling to use an "effective" method of contraception during the study and for up to 3 months after the use of study drug ceases.
* Patient has Î±-Fetoprotein more than 100ng/mL
* Patient has Hemoglobin <11g/dL (Male), 10g/dL (Female) or WBC count < 3,500/mm3 (PMN<1,500/mm3) or Platelet count <50,000/mm3
* Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2008-02; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBV DNA below 300copies/mL | at week 48

SECONDARY OUTCOMES:
The change of HBV DNA from the baseline | at week 24, 48
Proportion of patients with HBV DNA below LOD of RT-PCR | at week 24, 48
ALT normalization rate | at week 24, 48
Proportion of patients with viral breakthrough during 48-week treatment period | at week 24, 48

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Bundang
  - Seoul National University Hospital, Seoul